CLINICAL TRIAL: NCT05402592
Title: The Effect of Preoperative Oral Carbohydrate Administration on Postoperative Glucometabolic Response, Subjective Well-being and Quality of Life in Patients Undergoing Colorectal Surgery: A Randomized Prospective Trial
Brief Title: The Effect of Oral Carbohydrate Administration on Postoperative Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Cemile Celebi, Principal Investigator, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 22/12/2021-27/II
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Glucometabolic Response; Subjective Goodness; Life Quality
Keywords: colorectal cancer; carbonhydrate loading; carbonhydrate-rich drink; life quality; surgery; nursing care
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Water

STUDY DESIGN:
Intervention Model Description: Randomized Controlled prospective trial, double blind
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In the study, the participant, caregiver and outcome evaluator other than the researcher will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Patients will be given 800 ml of water by the blind caregiver until 24:00 at night before the surgery, and 400 ml of water 2-3 hours before the surgery in the morning.Blood samples for plasma glucose, plasma cortisol, and serum insulin levels will be drawn just before the morning dose, 40 minutes and 90 minutes after ingestion of the beverage, and during anesthesia induction. Gastric volume and pH will be evaluated within the first 10 minutes intraoperatively. Vital signs will be evaluated before, during and after surgery. To evaluate the biochemical parameters, blood samples will be taken again preoperatively and at the 6th and 24th hours postoperatively. Postoperative subjective well-being findings of the patients will be evaluated. The SF-36 quality of life scale will be applied to evaluate the quality of life of the patients on the 30th day after surgery.
  Interventions: Other: Water
- Carbonhydrate-rich drink (Experimental): Patients will be given 800 ml of carbohydrate-containing beverage until 24:00 at night before the surgery by the blind caregiver, and 400 ml of carbohydrate-containing beverage in the morning 2-3 hours before the surgery.Blood samples for plasma glucose, plasma cortisol, and serum insulin levels will be drawn just before the morning dose, 40 minutes and 90 minutes after ingestion of the beverage, and during anesthesia induction. Gastric volume and pH will be evaluated within the first 10 minutes intraoperatively. Vital signs will be evaluated before, during and after surgery. To evaluate the biochemical parameters, blood samples will be taken again preoperatively and at the 6th and 24th hours postoperatively. Postoperative subjective well-being findings of the patients will be evaluated. The SF-36 quality of life scale will be applied to evaluate the quality of life of the patients on the 30th day after surgery.
  Interventions: Dietary Supplement: Carbonhydrate rich drink

INTERVENTIONS:
Dietary Supplement: Carbonhydrate rich drink — It will be prepared by adding 50 g of carbohydrates to 1200 ml of water in total and will be given to the patients the night before the surgery and the morning of the surgery.
  Arms: Carbonhydrate-rich drink
Other: Water — A total of 1200 ml of water will be given to the patients the night before and the morning of the surgery.
  Arms: Control Group

SUMMARY:
Studies have shown that clear liquids containing carbohydrates are safe when given up to 2 hours before surgery and increase patient comfort before surgery. In the light of this information, this study aims to investigate the effects of preoperative oral carbohydrate administration on postoperative glucometabolic response, subjective well-being, quality of life, and surgical clinical outcomes in patients scheduled for colorectal surgery; planned as randomized-controlled, double-blind

DETAILED DESCRIPTION:
Fasting the night before surgery has been standard practice for patients undergoing elective surgery, with the expectation of minimizing the possibility of unwanted aspiration of gastric contents by emptying the stomach. Preoperative fasting increases perioperative insulin resistance (PIR) and patient discomfort. The surgery itself, especially a major procedure such as colorectal surgery, induces an endocrine and inflammatory stress response. PIR has an important role in the metabolic response to surgical trauma. PIR is a state of decreased glucose uptake in skeletal muscle and adipose tissue, with increased glucose secretion due to hepatic gluconeogenesis and hyperglycemia. A catabolic state occurs with glycogenolysis, muscle protein loss, and decreased storage of glycogen through lipolysis. The purpose of PIR is to provide energy and glycemic substrates to glucose-dependent tissues. PIR is an adaptive mechanism, but if left untreated, it can be harmful, increasing postoperative morbidity and mortality, and prolonging hospital stay . The level of insulin resistance formed; The duration of preoperative fasting, the type and duration of anesthesia and surgical technique, perioperative blood loss, and postoperative immobilization are related. Bilku et al. (2014) systematic review shows a significant reduction in insulin resistance in 6 of 7 randomized controlled trials. Wang et al. (2010) on 48 colorectal patients showed that insulin resistance was higher in patients who were conventionally fasted.As a result of recent advances in perioperative medicine, preoperative oral carbohydrate intake has been recommended as part of Advanced Post-Surgical Recovery (ERAS) protocols. The ERAS program was developed to facilitate postoperative recovery by reducing the stress response in colon surgery patients and includes various components of perioperative recommendations. ERAS recommends routine preoperative oral carbohydrate loading, especially for patients undergoing elective colon surgery. The aim of this is to reduce the stress response in the face of surgical trauma, to prevent complications, to shorten the recovery time, to minimize the hospital stay, to prevent postoperative morbidity and mortality. Preoperative oral liquid carbohydrate loading in the protocol; Before the planned surgical interventions, 800 ml of carbohydrate-rich liquid food is given to the individual until midnight, and 400 ml of liquid food 2-3 hours before the operation. The purpose of this application; In preoperative patients, metabolic satiety is achieved, insulin resistance, catabolism and blood glucose fluctuations are prevented.To avoid complications of pulmonary aspiration or laryngeal reflux, it is estimated that the volume of gastric contents should not exceed 200 mL prior to the surgical procedure. Several studies have detected a maximum mean gastric content of 120 mL, ranging from 10-30 mL after a clear liquid diet up to 2 hours before surgery. Bilku et al. (2014) found that gastric content volume and pH were nearly identical between conventional fasting and shortened 2-hour fasting. Both clear liquids and carbohydrate solutions were drained in approximately 90 minutes. The authors concluded that there was no increased risk of aspiration or regurgitation in patients with a shortened 2-hour fast. Yagci et al. (2008) also concluded in a study involving 70 patients who had undergone cholecystectomy or thyroidectomy, that administration of carbohydrate drinks 2 hours before did not change gastric pH or content volume.Traditional fasting puts the patient in a catabolic state and intensifies the patient's response to trauma. Surgical delay may increase this effect. Fluids containing complex carbohydrates (usually around 12% carbohydrates, predominantly in the form of maltodextrin to limit osmolality and prevent delayed gastric emptying) given 2-3 hours before the procedure produce a more anabolic state, stimulate postprandial glycemia, reduce glycogen loss, and increase by skeletal muscle Hyperglycemia is controlled by glucose uptake.It has been reported that perioperative thirst, hunger, weakness, fatigue and anxiety improve with the reduction of fasting time and the use of carbohydrate-containing fluids. Hausel et al. (2005) found that preoperatively, the carbohydrate group was less hungry and anxious compared to the placebo and fasting groups, and the feeling of thirst decreased in both carbohydrate drink and placebo groups. It was determined that the carbohydrate group also experienced less fatigue and discomfort. A remarkable inability to concentrate and an increase in weakness, hunger, and thirst were reported in the fasted group. In a study conducted in our country, it was reported that 47.1% of the nurses did not take any action for patients who had prolonged surgery. In the study conducted by Bopp et al. (2011), patients who were fasted after midnight before the operation and who were given a carbohydrate solution two hours before the operation were compared, it was reported that the intervention group did not feel hunger or thirst before the operation, and that their post-operative satisfaction and comfort increased.Postoperative nausea-vomiting (ASBK), which is thought to be due to surgical stress, prolonged fasting time, and anesthetic agents and is among the most common complications after surgery, is 30-45% in risk group, especially in individuals at risk for gastric problems and in major surgical interventions. in individuals, it is seen at rates as high as 80%. It is stated that approximately one third of all patients undergoing surgical intervention experience ASBK. ASBK causes discomfort, anxiety, and indirectly or directly an increase in pain in the individual. In some studies on the effect of carbohydrate fluids on postoperative nausea and vomiting, it is stated that oral carbohydrate solution administration before surgery has positive effects on postoperative nausea and vomiting. It is thought that this positive effect occurs as a result of the helper effect of carbohydrate, which provides a source for glucose metabolism, in the regulation of blood glucose levels.It is emphasized that preoperative oral carbohydrate intake can reduce hospitalization due to its positive effects on insulin resistance and gastrointestinal symptoms. Awad et al. (2013) reported that it significantly reduced hospitalization in patients undergoing major abdominal surgery. Mathur et al. (2010) also determined that intestinal function returned earlier in the carbohydrate group, although there was no statistical significance. Noblett et al. (2006) found in their randomized controlled trial that hospitalizations were reduced in the carbohydrate group and that the return of gastrointestinal function was accelerated.Studies have shown that clear liquids containing carbohydrates are safe when given up to 2 hours before surgery and increase patient comfort before surgery. In the light of this information, this study aims to investigate the effects of preoperative oral carbohydrate administration on postoperative glucometabolic response, subjective well-being, quality of life, and surgical clinical outcomes in patients scheduled for colorectal surgery; planned as randomized-controlled, double-blind

ELIGIBILITY:
Inclusion Criteria:

* Those who agree to participate in the study, have the ability to make decisions,
* Patients aged 18 and over,
* Patients who will undergo colorectal surgery,
* Patients with ASA I-II-III

Exclusion Criteria:

* Diabetes diagnosis,
* Patient with oral feeding problem
* Gastric emptying is delayed,
* Diagnosed with gastroesophageal reflux,
* Having a diagnosis of hiatal hernia,
* Severe liver or kidney failure,
* Having symptoms of glucometabolic imbalance,
* Emergency patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
glucometabolic well-being | within postoperative 24 hours
  To reduce insulin resistance, HOMA-IR value is expected to be below 2.5 mg/dL. HOMA-IR=Fasting Plasma Glucose (mmol/L) × Fasting insulin (mU/L) / 22.5
Subjective well-being | within postoperative 24 hours
  Low scores on the numerical pain scale of subjective data such as pain, thirst, hunger, dry mouth, pain at rest, pain with mobilization, nausea, vomiting, weakness, and anxiety indicate subjective well-being.
Shorter Length Of Hospitalization | within postoperative 24 hours
  Total amount of days spent in hospital

SECONDARY OUTCOMES:
Assessment of postoperative pain | At moment 0, 2, 4, 8 12 and 24 hours after surgery
  NRS scale (from 0 to 10, 0 is no pain, 10 is maximum pain)
Presence/Absence of nausea | At moment 0, 2, 4, 8 12 and 24 hours after surgery
  NRS scale (from 0 to 10, 0 is no nausea, 10 is maximum nausea)
Presence/Absence of vomiting | At moment 0, 2, 4, 8 12 and 24 hours after surgery
  NRS scale (from 0 to 10, 0 is no vomiting, 10 is maximum vomiting)
Time to hunger | At moment 0, 2, 4, 8 12 and 24 hours after surgery
  NRS scale (from 0 to 10, 0 is no hunger, 10 is maximum hunger)
mouth dry | At moment 0, 2, 4, 8 12 and 24 hours after surgery
  NRS scale (from 0 to 10, 0 is no mouth dry, 10 is maximum mouth dry)
Time to flatus | Up to 4 weeks after surgery
  Hours elapsed to event
Time to bowel movement | Up to 4 weeks after surgery
  Hours elapsed to event
Higher quality of life on the 30th day after surgery in patients given a carbohydrate-rich beverage before surgery | Up to 4 weeks after surgery
  Patients given a carbohydrate-rich beverage preoperatively are expected to score high on the SF-36 scale on the 30th day after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Urkan, Assoc. Prof., Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla Sıtkı Koçman University, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All data of the study will be shared with the researchers who request it.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Indefinitely
Access Criteria: Research, meta-analysis

REFERENCES:
- [Background] Awad S, Varadhan KK, Ljungqvist O, Lobo DN. A meta-analysis of randomised controlled trials on preoperative oral carbohydrate treatment in elective surgery. Clin Nutr. 2013 Feb;32(1):34-44. doi: 10.1016/j.clnu.2012.10.011. Epub 2012 Nov 7. PMID 23200124
- [Background] Bilku DK, Dennison AR, Hall TC, Metcalfe MS, Garcea G. Role of preoperative carbohydrate loading: a systematic review. Ann R Coll Surg Engl. 2014 Jan;96(1):15-22. doi: 10.1308/003588414X13824511650614. PMID 24417824
- [Background] Bopp C, Hofer S, Klein A, Weigand MA, Martin E, Gust R. A liberal preoperative fasting regimen improves patient comfort and satisfaction with anesthesia care in day-stay minor surgery. Minerva Anestesiol. 2011 Jul;77(7):680-6. Epub 2009 Feb 4. PMID 19190563
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Hausel J, Nygren J, Thorell A, Lagerkranser M, Ljungqvist O. Randomized clinical trial of the effects of oral preoperative carbohydrates on postoperative nausea and vomiting after laparoscopic cholecystectomy. Br J Surg. 2005 Apr;92(4):415-21. doi: 10.1002/bjs.4901. PMID 15739210
- [Background] Hubner M, Addor V, Slieker J, Griesser AC, Lecureux E, Blanc C, Demartines N. The impact of an enhanced recovery pathway on nursing workload: A retrospective cohort study. Int J Surg. 2015 Dec;24(Pt A):45-50. doi: 10.1016/j.ijsu.2015.10.025. Epub 2015 Oct 30. PMID 26523495
- [Background] Jones C, Badger SA, Hannon R. The role of carbohydrate drinks in pre-operative nutrition for elective colorectal surgery. Ann R Coll Surg Engl. 2011 Oct;93(7):504-7. doi: 10.1308/147870811X13137608455136. PMID 22004631
- [Background] Li L, Wang Z, Ying X, Tian J, Sun T, Yi K, Zhang P, Jing Z, Yang K. Preoperative carbohydrate loading for elective surgery: a systematic review and meta-analysis. Surg Today. 2012 Jul;42(7):613-24. doi: 10.1007/s00595-012-0188-7. Epub 2012 May 13. PMID 22581289
- [Background] Ljungqvist O. Jonathan E. Rhoads lecture 2011: Insulin resistance and enhanced recovery after surgery. JPEN J Parenter Enteral Nutr. 2012 Jul;36(4):389-98. doi: 10.1177/0148607112445580. Epub 2012 May 10. PMID 22577121
- [Background] Ljungqvist O, Soreide E. Preoperative fasting. Br J Surg. 2003 Apr;90(4):400-6. doi: 10.1002/bjs.4066. PMID 12673740
- [Background] Mathur S, Plank LD, McCall JL, Shapkov P, McIlroy K, Gillanders LK, Merrie AE, Torrie JJ, Pugh F, Koea JB, Bissett IP, Parry BR. Randomized controlled trial of preoperative oral carbohydrate treatment in major abdominal surgery. Br J Surg. 2010 Apr;97(4):485-94. doi: 10.1002/bjs.7026. PMID 20205227
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Noblett SE, Watson DS, Huong H, Davison B, Hainsworth PJ, Horgan AF. Pre-operative oral carbohydrate loading in colorectal surgery: a randomized controlled trial. Colorectal Dis. 2006 Sep;8(7):563-9. doi: 10.1111/j.1463-1318.2006.00965.x. PMID 16919107
- [Background] Pimenta GP, de Aguilar-Nascimento JE. Prolonged preoperative fasting in elective surgical patients: why should we reduce it? Nutr Clin Pract. 2014 Feb;29(1):22-8. doi: 10.1177/0884533613514277. Epub 2013 Dec 11. PMID 24336400
- [Background] Pogatschnik C, Steiger E. Review of Preoperative Carbohydrate Loading. Nutr Clin Pract. 2015 Oct;30(5):660-4. doi: 10.1177/0884533615594013. Epub 2015 Jul 21. PMID 26197803
- [Background] Smith I, Kranke P, Murat I, Smith A, O'Sullivan G, Soreide E, Spies C, in't Veld B; European Society of Anaesthesiology. Perioperative fasting in adults and children: guidelines from the European Society of Anaesthesiology. Eur J Anaesthesiol. 2011 Aug;28(8):556-69. doi: 10.1097/EJA.0b013e3283495ba1. PMID 21712716
- [Background] Smith HS, Smith EJ, Smith BR. Postoperative nausea and vomiting. Ann Palliat Med. 2012 Jul;1(2):94-102. doi: 10.3978/j.issn.2224-5820.2012.07.05. PMID 25841469
- [Background] Wang ZG, Wang Q, Wang WJ, Qin HL. Randomized clinical trial to compare the effects of preoperative oral carbohydrate versus placebo on insulin resistance after colorectal surgery. Br J Surg. 2010 Mar;97(3):317-27. doi: 10.1002/bjs.6963. PMID 20101593
- [Background] Yagci G, Can MF, Ozturk E, Dag B, Ozgurtas T, Cosar A, Tufan T. Effects of preoperative carbohydrate loading on glucose metabolism and gastric contents in patients undergoing moderate surgery: a randomized, controlled trial. Nutrition. 2008 Mar;24(3):212-6. doi: 10.1016/j.nut.2007.11.003. Epub 2007 Dec 21. PMID 18096368
- [Result] Akbarzadeh M, Eftekhari MH, Shafa M, Alipour S, Hassanzadeh J. Effects of a New Metabolic Conditioning Supplement on Perioperative Metabolic Stress and Clinical Outcomes: A Randomized, Placebo-Controlled Trial. Iran Red Crescent Med J. 2016 Jan 9;18(1):e26207. doi: 10.5812/ircmj.26207. eCollection 2016 Jan. PMID 26889394
- [Derived] Urkan M, Celebi C, Meral UM, Cavdar I. The effect of preoperative oral carbohydrate administration on postoperative glucometabolic response, subjective well being and quality of life in patients undergoing colorectal surgery: a randomized controlled double-blind study. BMC Surg. 2025 Aug 20;25(1):376. doi: 10.1186/s12893-025-03093-3. PMID 40830867
- See also: 8. Çilingir D, Candaş B. Cerrahi sonrası hızlandırılmış iyileşme protokolü ve hemşirenin rolü. Journal of Anatolia Nursing and Health Sciences 2017;20(2):137-143. — https://dergipark.org.tr/tr/pub/ataunihem/issue/31359/342629
- See also: 7. Çakır SK, Van Giersbergen MY, Umar DÇ. Cerrahi hemşirelerinin ameliyat öncesi aç kalma ile ilgili uygulama ve bilgi düzeyi. Ege Üniversitesi Hemşirelik Fakültesi Dergisi. 2018;34(1):26-35. — https://dergipark.org.tr/tr/pub/egehemsire/issue/36787/301646
- See also: 3. Aygin, D. (2016). Bulantı ve Kusma. Yoğun Bakım Hemşireliği Dergisi, 20(1), 44-56. — https://dergipark.org.tr/tr/pub/ybhd/issue/26500/278837

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT05402592/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT05402592/ICF_001.pdf